CLINICAL TRIAL: NCT03318549
Title: Brain-Computer Interface (BCI) and Evaluation of Visual and Task Performance in Subjects With Eye Diseases
Brief Title: BCI and Evaluation of Visual and Task Performance in Subjects With Eye Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Felipe Andrade Medeiros, Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20240020; Pro00088016 (Other: Duke University); R01EY029885 (NIH)
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Glaucoma; Macular Degeneration; Glaucoma Suspect; Optic Neuropathy; Retinal Degeneration; Visual Pathway Disorder
Keywords: virtual reality; glaucoma; age related macular degeneration; quality of life; visual field; optical coherence tomography; brain-computer interface
MeSH Terms: conditions — Glaucoma; Macular Degeneration; Ocular Hypertension; Optic Nerve Diseases; Retinal Degeneration | interventions — Brain-Computer Interfaces

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Glaucoma group (Other): Patients with diagnosed glaucoma will be in the group for up to 5 years.
  Interventions: Diagnostic Test: Visual Performance tests; Device: Brain-computer interface
- Suspicious of having glaucoma group (Other): Patients with suspicious of having glaucoma will be in the group for up to 5 years.
  Interventions: Diagnostic Test: Visual Performance tests; Device: Brain-computer interface
- Non-glaucomatous optic neuropathies group (Other): Patients with optic neuropathies that do not look glaucomatous-like will be in the group for up to 5 years.
  Interventions: Diagnostic Test: Visual Performance tests
- Age-related macular degeneration (AMD) group (Other): Patients with diagnosed age-related macular degeneration will be in the group for up to 5 years.
  Interventions: Diagnostic Test: Visual Performance tests
- Retinal degenerations group (Other): Patients with other retinal degenerations excluding AMD will be in the group for up to 5 years.
  Interventions: Diagnostic Test: Visual Performance tests
- Other diseases of visual pathways group (Other): Other diseases of the visual pathway not included in the previous groups will be in the group for up to 5 years.
  Interventions: Diagnostic Test: Visual Performance tests
- Healthy control group (Other): Patients labeled as healthy controls for not having any other eye diseases that would be included on the other groups will be in the group for up to 5 years.
  Interventions: Diagnostic Test: Visual Performance tests; Device: Brain-computer interface

INTERVENTIONS:
Diagnostic Test: Visual Performance tests — Participants came to the clinic in person for 2 hours for visual performance tests once every 6 months for up to 5 years. These tests included virtual reality tests and tests on a computer screen to investigate performance during simulated daily life activities, such as driving, situations of low contrast and glare.
Device: Brain-computer interface — The brain-computer interface (BCI) consists of a modified virtual reality goggle integrated with wireless no-prep electroencephalogram (EEG). The portable BCI is able to objectively measure multifocal steadystate visual evoked potentials in response to brain stimulation through presentation of visual stimuli in the goggle. The test is done in person and may take up to 30 minutes, once every 6 months for up to 5 years.
  Arms: Glaucoma group; Healthy control group; Suspicious of having glaucoma group

SUMMARY:
The purpose of this research study is to better understand the impact of visual impairment caused by different eye diseases on the ability to perform daily activities and compare it to that in patients without eye diseases.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between the ages of 18 and 90 years old;
* Both males and females will be included.
* Be able and willing to provide signed informed consent and follow study instructions

Exclusion Criteria:

* Subjects will be excluded if they present with any systemic conditions that in the opinion of the Principal Investigator may prevent them from completing the tests.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe A Medeiros, MD, PhD, Principal Investigator — University of Miami; Henry Tseng, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Bascom Palmer Eye Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No patients were enrolled during the study period for groups: Non-glaucomatous optic neuropathies group; Age-related macular degeneration (AMD) group; Retinal degenerations group; Other diseases of visual pathways group.
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | Healthy Control Group | Glaucoma Group | Suspicious of Having Glaucoma Group | Non-glaucomatous Optic Neuropathies Group | Age-related Macular Degeneration (AMD) Group | Retinal Degenerations Group | Other Diseases of Visual Pathways Group
Started | 14; 28 eyes | 89; 178 eyes | 12; 24 eyes | 0; 0 eyes | 0; 0 eyes | 0; 0 eyes | 0; 0 eyes
Completed | 9; 18 eyes | 63; 126 eyes | 6; 12 eyes | 0; 0 eyes | 0; 0 eyes | 0; 0 eyes | 0; 0 eyes
Not Completed | 5; 10 eyes | 26; 52 eyes | 6; 12 eyes | 0; 0 eyes | 0; 0 eyes | 0; 0 eyes | 0; 0 eyes
Not completed — Withdrawal by Subject | 5 | 19 | 2 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 4 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 3 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patients were enrolled during the study period for groups: Non-glaucomatous optic neuropathies group; Age-related macular degeneration (AMD) group; Retinal degenerations group; Other diseases of visual pathways group.
Units Other Than Participants: eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Control Group | Glaucoma Group | Suspicious of Having Glaucoma Group | Non-glaucomatous Optic Neuropathies Group | Age-related Macular Degeneration (AMD) Group | Retinal Degenerations Group | Other Diseases of Visual Pathways Group | Total
Number analyzed (Participants) | 14 | 89 | 12 | 0 | 0 | 0 | 0 | 115
Number analyzed (eyes) | 28 | 178 | 24 | 0 | 0 | 0 | 0 | 230
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (4.2) | 67.7 (9.7) | 67.2 (10.0) |  |  |  |  | 68.2 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 52 | 4 |  |  |  |  | 64
  Male | 6 | 37 | 8 |  |  |  |  | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 |  |  |  |  | 2
  Not Hispanic or Latino | 14 | 87 | 12 |  |  |  |  | 113
  Unknown or Not Reported | 0 | 0 | 0 |  |  |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 |  |  |  |  | 0
  Asian | 0 | 3 | 1 |  |  |  |  | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  |  |  |  | 0
  Black or African American | 1 | 26 | 4 |  |  |  |  | 31
  White | 13 | 58 | 7 |  |  |  |  | 78
  More than one race | 0 | 0 | 0 |  |  |  |  | 0
  Unknown or Not Reported | 0 | 2 | 0 |  |  |  |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Visual Impairment Measured by Visual Functioning Test
Description: The study team will evaluate visual impairment through a composite score of visual functioning test, ranging from 0 to 100, with lower scores indicating worse visual impairment.
Time Frame: 4.5 years
Population: Two subjects with eyes with visual function tests with low reliability scores were excluded from the analysis. Monocular patients were included. No patients were enrolled during the study period for groups: Non-glaucomatous optic neuropathies group; Age-related macular degeneration (AMD) group; Retinal degenerations group; Other diseases of visual pathways group.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Healthy Control Group | Glaucoma Group | Suspicious of Having Glaucoma Group | Non-glaucomatous Optic Neuropathies Group | Age-related Macular Degeneration (AMD) Group | Retinal Degenerations Group | Other Diseases of Visual Pathways Group
Number analyzed (Participants) | 14 | 88 | 11 | 0 | 0 | 0 | 0
Number analyzed (eyes) | 28 | 170 | 20 | 0 | 0 | 0 | 0
score on a scale | 80.6 (5.3) | 74.2 (13.0) | 81.1 (10.4) |  |  |  |
Statistical Analysis 1: Comparison: Healthy Control Group vs Glaucoma Group; Test type: Other; p = 0.011, t-test, 2 sided
Statistical Analysis 2: Comparison: Glaucoma Group vs Suspicious of Having Glaucoma Group; Test type: Other; p = 0.022, t-test, 2 sided

2. Primary Outcome: Number of Eyes Showing Progression
Description: The number of eyes showing progression (expressed in percentage) will be compared between the home-based Brain-computer interface (BCI) testing and standard clinical testing (standard automated perimetry, SAP)
Time Frame: 4.5 years
Population: Two subjects with eyes with visual function tests with low reliability scores were excluded from the analysis. Monocular patients were included. No patients were enrolled during the study period for groups: Non-glaucomatous optic neuropathies group; Age-related macular degeneration (AMD) group; Retinal degenerations group; Other diseases of visual pathways group. Healthy Control Group Arm, participants in this Arm were not assessed for this endpoint, and therefore, no data were collected.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Healthy Control Group | Glaucoma Group | Suspicious of Having Glaucoma Group | Non-glaucomatous Optic Neuropathies Group | Age-related Macular Degeneration (AMD) Group | Retinal Degenerations Group | Other Diseases of Visual Pathways Group
Number analyzed (Participants) | 0 | 88 | 11 | 0 | 0 | 0 | 0
Number analyzed (eyes) | 0 | 170 | 20 | 0 | 0 | 0 | 0
eyes
  Progression by BCI only |  | 33 | 7 |  |  |  |
  Progression by SAP only |  | 26 | 0 |  |  |  |
  Progression by BCI and SAP |  | 15 | 2 |  |  |  |
  No progression |  | 96 | 11 |  |  |  |
Statistical Analysis 1: Comparison: Glaucoma Group vs Suspicious of Having Glaucoma Group; Test type: Other; p = 0.303, Chi-squared

3. Primary Outcome: Time to Detect Progression Measured in Years
Description: The time to detect progression (years) will be compared between the home-based Brain-computer interface testing and standard clinical testing (standard automated perimetry).
Time Frame: 4.5 years
Population: Monocular patients were included. No patients were enrolled during the study period for groups: Non-glaucomatous optic neuropathies group; Age-related macular degeneration (AMD) group; Retinal degenerations group; Other diseases of visual pathways group. Healthy Control Group Arm, participants in this Arm were not assessed for this endpoint, and therefore, no data were collected. Data collected for progressing eyes with a minimum of 1.5 years of follow-up.
Measure: Mean (Standard Deviation); unit: years
Units Other Than Participants: eyes
Arm/Group | Healthy Control Group | Glaucoma Group | Suspicious of Having Glaucoma Group | Non-glaucomatous Optic Neuropathies Group | Age-related Macular Degeneration (AMD) Group | Retinal Degenerations Group | Other Diseases of Visual Pathways Group
Number analyzed (Participants) | 0 | 11 | 1 | 0 | 0 | 0 | 0
Number analyzed (eyes) | 0 | 17 | 2 | 0 | 0 | 0 | 0
years
  SAP |  | 3.3 (1.3) | 2.9 (0.0) |  |  |  |
  BCI |  | 2.7 (1.5) | 2.9 (0.0) |  |  |  |

4. Secondary Outcome: Standard Automated Perimetry Will be Assessed by the C-index
Description: c-index will be calculated by the proportion of concordant pairs divided by the total number of possible evaluation pairs for progression. c-index is unitless.
Time Frame: 4.5 years
Population: Two subjects with eyes with visual function tests with low reliability scores were excluded from the analysis. Monocular patients were included. No patients were enrolled during the study period for groups: Non-glaucomatous optic neuropathies group; Age-related macular degeneration (AMD) group; Retinal degenerations group; Other diseases of visual pathways group. Healthy Control Group Arm: participants in this Arm were not assessed for this endpoint, and therefore, no data were collected.
Measure: Number; unit: unitless
Units Other Than Participants: eyes
Arm/Group | Healthy Control Group | Glaucoma Group | Suspicious of Having Glaucoma Group | Non-glaucomatous Optic Neuropathies Group | Age-related Macular Degeneration (AMD) Group | Retinal Degenerations Group | Other Diseases of Visual Pathways Group
Number analyzed (Participants) | 0 | 88 | 11 | 0 | 0 | 0 | 0
Number analyzed (eyes) | 0 | 170 | 20 | 0 | 0 | 0 | 0
unitless |  | .652 | .667 |  |  |  |

5. Secondary Outcome: Patient-reported Quality of Life as Measured by the National Eye Institute (NEI) Visual Function Questionnaire (VFQ) 25
Description: The scores on the NEI VFQ-25 subscale ranges from 0 to 100, with a higher score indicating greater functioning.
Time Frame: 4.5 years
Population: Subjects with questionnaires with incomplete responses were excluded from the analysis. No patients were enrolled during the study period for groups: Non-glaucomatous optic neuropathies group; Age-related macular degeneration (AMD) group; Retinal degenerations group; Other diseases of visual pathways group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Control Group | Glaucoma Group | Suspicious of Having Glaucoma Group | Non-glaucomatous Optic Neuropathies Group | Age-related Macular Degeneration (AMD) Group | Retinal Degenerations Group | Other Diseases of Visual Pathways Group
Number analyzed (Participants) | 13 | 87 | 11 | 0 | 0 | 0 | 0
score on a scale | 95.2 (6.1) | 91.3 (8.9) | 92.6 (5.1) |  |  |  |
Statistical Analysis 1: Comparison: Healthy Control Group vs Glaucoma Group; Test type: Other; p = 0.132, t-test, 2 sided
Statistical Analysis 2: Comparison: Glaucoma Group vs Suspicious of Having Glaucoma Group; Test type: Other; p = 0.647, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 4.5 years
Description: No patients were enrolled during the study period for groups: Non-glaucomatous optic neuropathies group; Age-related macular degeneration (AMD) group; Retinal degenerations group; Other diseases of visual pathways group.
Arm/Group | Healthy Control Group | Glaucoma Group | Suspicious of Having Glaucoma Group | Non-glaucomatous Optic Neuropathies Group | Age-related Macular Degeneration (AMD) Group | Retinal Degenerations Group | Other Diseases of Visual Pathways Group
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/89 | 0/12 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/89 | 0/12 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/14 | 0/89 | 0/12 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
No patients were enrolled during the study period for groups: Non-glaucomatous optic neuropathies group; Age-related macular degeneration (AMD) group; Retinal degenerations group; Other diseases of visual pathways group. A limited number of patients reached the 5-year follow-up mark, which did not provide enough power for progression analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT03318549/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT03318549/ICF_001.pdf